CLINICAL TRIAL: NCT01446601
Title: Pivotal Study of the Apnex Medical™ Hypoglossal Nerve Stimulation (HGNS) System to Treat Obstructive Sleep Apnea
Brief Title: Apnex Clinical Study of the Hypoglossal Nerve Stimulation (HGNS®) System to Treat Obstructive Sleep Apnea
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Apnex Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLP-005; IDE #G090014 (Other: FDA)
Record Dates: First submitted 2011-09-02; First posted 2011-10-05 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2011-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: Apnea; OSA; Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Hypoglossal Nerve Stimulation; Sleep Disorders; Tongue
MeSH Terms: conditions — Sleep Apnea, Obstructive; Apnea; Sleep Apnea Syndromes; Sleep Wake Disorders | interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): The Treatment Arm is implanted with the HGNS System and therapy is turned on at 1 month post-implant.
  Interventions: Device: Hypoglossal Nerve Stimulation (HGNS) System (Apnex Medical )
- Control (Other): The Control Arm is implanted with the HGNS System and therapy is turned on at 7 months post-implant.
  Interventions: Device: Hypoglossal Nerve Stimulation (HGNS) System (Apnex Medical )

INTERVENTIONS:
Device: Hypoglossal Nerve Stimulation (HGNS) System (Apnex Medical ) — The HGNS System in an investigational device that includes three implantable components: a neurostimulator, a stimulation lead, and a respiration sensing lead. The HGNS System is designed to activate the muscles in the upper airway to help keep the airway open during sleep. The HGNS System is intended for the treatment of moderate to severe OSA in individuals that have failed or do not tolerate positive airway pressure (PAP) therapy.

SUMMARY:
The purpose of this study is to evaluate the benefits and risks of hypoglossal nerve stimulation with the Apnex Medical Hypoglossal Nerve Stimulation (HGNS) System as a potential therapeutic option for individuals with moderate to severe Obstructive Sleep Apnea (OSA) that have failed or do not tolerate positive airway pressure (PAP) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 80 years
* Body mass index (BMI) ≤ 35 kg/m²
* Previously diagnosed with Moderate to severe OSA
* Individual has failed or does not tolerate PAP therapy

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Reduction in OSA Severity | from Baseline to 6 Months
  The proportion of subjects that experience clinically meaningful improvement in AH1 (reduction >50% and AHI <20) and ODI 4% (reduction >= 25% or ODI 4% <5)from Baseline to 6 Months will be significantly greater in the Treatment Group compared to the Control Group
Long-term Reduction in OSA Severity | 12 months
  The proportion of subjects in the Treatment Group that experience clinically relevant improvement in AHI (reduction >50% and AHI <20) and ODI 4% (reduction >=25% or ODI 4% <5 at 12 months compared to Baseline.
Safety Analysis | 12 months
  Description of all adverse events

CONTACTS AND LOCATIONS:
Locations (14):
- United States (12):
  - MidAmerica Neuroscience Research Institute, Lenexa, Kansas
  - Veritas Clinical Specialties, Topeka, Kansas
  - Kentucky Research Group, Louisville, Kentucky
  - The Center for Sleep and Wake Disorders, Chevy Chase, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - St. Lukes Hospital, St Louis, Missouri
  - Clinilabs, New York, New York
  - Wilmington Medical Research, Wilmington, North Carolina
  - Community Research, Cincinnati, Ohio
  - Sleep Med of South Carolina, Columbia, South Carolina
  - Sleep Therapy and Research Center, San Antonio, Texas
- Australia (2):
  - Westmead Hospital, Sydney, New South Wales
  - IBAS, The Austin Hospital, Melbourne, Victoria